CLINICAL TRIAL: NCT02279355
Title: Peri-operative Risk Factors for Postoperative Pressure Ulcer in Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0323
Record Dates: First submitted 2014-10-13; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Postoperative Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pressure ulcer group: Patient who developing pressure ulcer categorized as stage more than II after surgery
- Control group: Patients has identical values on the matching factors such as age, sex and surgical procedures of control group

SUMMARY:
The aim of this retrospective study is to overall evaluate and validate preoperative and intra-operative risk factors for postoperative pressure ulcers in critically ill postoperative patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients in ICU with a greater than 48 hours
* Underwent a surgical procedures,
* Absence of pressure ulcer present at admission to the ICU and developed a stage II or higher pressure ulcer, deep tissue injury, or unstageable ulcer, as defined by the pressure ulcer staging guidelines of the National Pressure Ulcer Advisory Panel.

Exclusion Criteria:

* Patients will be excluded from the study if they had been diagnosed with pressure ulcer before the surgery
* Pediatric patients

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total about 130 adult surgical patients underwent surgical procedures and admitted in intensive care unit (ICU) using electronic documentation applications from Jan 2012 through Dec 2013.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
independent preoperative risk factors | up to1 month after surgery
  Postoperative new-onset pressure ulcers were identified from nursing documentation in the patient's electrical medical record within 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Na, MD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute Yonsei University College of Medicine